CLINICAL TRIAL: NCT04451421
Title: Effects of Standing at Different Angles on Transpulmonary Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: transpulmonary pressure
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standing Angle (Experimental): Assist the electric hospital bed to conduct different Angle standing training, starting from 20 degrees, every five minutes to rise 5 degrees, the maximum rise to 80 degrees
  Interventions: Behavioral: Change of standing Angle

INTERVENTIONS:
Behavioral: Change of standing Angle — Change the patient's standing Angle by using an electric bed

SUMMARY:
Effects of standing at different angles on transpulmonary pressure

DETAILED DESCRIPTION:
Objective: To study the effect of different standing angles on cross-lung pressure.Background: Long-term bed rest in ICU patients leads to upward movement of diaphragm and increased intrathoracic pressure in mechanically ventilated patients, resulting in lower cross-lung pressure. If the end-expiratory cross-lung pressure is negative, lung tissue compression and atelectasis will occur.Standing can lower the diaphragm, improve the pressure across the lungs, and improve ventilation.Selection methods: patients with invasive mechanical ventilation in the ICU, on the premise of stable hemodynamics, with the aid of electric bed training in standing in different angles, start from 20 degrees, 5 degrees up every five minutes, the largest up to 80 degrees, each Angle across the pulmonary pressure, die cavity ratio, tidal volume and breathe out carbon dioxide at the end of the record, and record whether low blood pressure, an accident in the process of take off the tube and other adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* The age is ≥ 18 years old;
* the hemodynamics is stable;
* 50 < heart rate < 120 beats / min ;
* 90 < systolic blood pressure < 200mmHg ;
* 55 < mean arterial pressure < 120mmHg;
* do not increase the dose of pressor drugs for at least 2 hours;
* intracranial pressure is stable and there are no seizures within 24 hours;
* the respiratory state is stable;
* the patient's finger pulse oxygen saturation ≥ 88%;
* 10 < respiratory frequency < 35 beats / min.

Exclusion Criteria:

* Pregnancy;
* acute cardio-cerebrovascular events;
* spinal or limb fractures;
* active bleeding.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
transpulmonary pressure | 5 minutes
  End-expiratory pressure across the lungs is recommended at 0-5cmH2O.
Esophageal pressure | 5 minutes
  The change in esophageal pressure represents the degree of inspiratory effort.The greater the variation, the harder the inhale.
Dead space rate | 5 minutes
  the smaller，the better
tidal volume | 5 minutes
  Standard tidal volume: standard weight based on height, 6 to 8ml per kg body weight
partial pressure of carbon dioxide in endexpiratory gas | 5 minutes
  The smaller the difference between pCO2 and arterial blood gas, the better

SECONDARY OUTCOMES:
adverse reaction | an hour
  hypotension、Accident to take off the tube、Drop of bed，Record the number of times it happens.The more it happens, the less safe it is.

CONTACTS AND LOCATIONS:
Overall Officials: xin li xie, Ph.D., Principal Investigator — The First Medical Center of PLA General Hospital